CLINICAL TRIAL: NCT04355728
Title: Umbilical Cord-derived Mesenchymal Stem Cells for COVID-19 Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Use of UC-MSCs for COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Camillo Ricordi (Other)
Responsible Party: Sponsor-Investigator, Camillo Ricordi, Professor of Surgery and Chief, Division of Cellular Transplantation, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200671; 20200370 (Other: Secondary Protocol ID)
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Corona Virus Infection; ARDS; ARDS, Human; Acute Respiratory Distress Syndrome; COVID-19
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: The trial has two groups, each with 12 subjects (n=24). All eligible subjects will be randomized to either the treatment group or standard of care, and randomization will be stratified by ARDS severity.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinding Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UC-MSCs Group (Experimental): Participants in this group will be treated with two infusions of UC-MCSs along with heparin (blood thinner) in addition to standard of care treatment. The first infusion will be administered within 24 hours of study enrollment and the second infusion will be administered within 72 hours of study enrollment.
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells + Heparin along with best supportive care.
- Control Group (Placebo Comparator): Participants in this group will be treated with two infusions of vehicle along with heparin (blood thinner) in addition to standard of care treatment. The first infusion will be administered within 24 hours of study enrollment and the second infusion will be administered within 72 hours of study enrollment.
  Interventions: Other: Vehicle + Heparin along with best supportive care

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells + Heparin along with best supportive care. — UC-MSC will be administered at 100x10^6 cells/infusion administered intravenously in addition to the standard of care treatment.
  Arms: UC-MSCs Group
Other: Vehicle + Heparin along with best supportive care — Best supportive care treatment per the treating hospital protocol.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to learn about the safety and efficacy of human umbilical cord derived Mesenchymal Stem Cells (UC-MSC) for treatment of COVID-19 Patients with Severe Complications of Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS).

ELIGIBILITY:
Inclusion Criteria:

Patients >/= 18 years old diagnosed with COVID-19 (as evaluated by PCR test confirming infection with SARS-CoV-2) will be eligible for inclusion if they meet all of the below criteria. Inclusion criteria must all be present within a 24-hour time period at the time of enrollment:

1. Patient currently hospitalized
2. Aged ≥ 18 years
3. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent
4. Peripheral capillary oxygen saturation (SpO2) ≤ 94% at room air, or requiring supplemental oxygen at screening
5. PaO2/FiO2 ratio < 300 mmHg
6. Bilateral infiltrates on frontal chest radiograph or bilateral ground glass opacities on a chest CT scan
7. Hypoxemia requiring an increase in the fraction of inspired oxygen (FiO2) of ≥ 20% AND an increase in positive end-expiratory airway pressure (PEEP) level of 5 cm H2O or more to maintain transcutaneous oxygen saturations in the target range of 88-95%, or requirement for escalation from oxygen therapy to invasive mechanical ventilation

Exclusion Criteria:

1. PaO2/FiO2 ≥ 300 at the time of enrollment
2. A previous MSC infusion not related to this trial
3. History of Pulmonary Hypertension (WHO Class III/IV)
4. History of left atrial hypertension or decompensated left heart failure.
5. Pregnant or lactating patient
6. Unstable arrhythmia
7. Patients with previous lung transplant
8. Patients currently receiving chronic dialysis
9. Patients currently receiving Extracorporeal Membrane Oxygenation (ECMO)
10. Presence of any active malignancy (except non-melanoma skin cancer)
11. Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
12. Moderate to severe liver disease (AST and ALT >5 X ULN)
13. Severe chronic respiratory disease with a PaCO2 > 50 mm Hg or the use of home oxygen
14. Baseline QT prolongation
15. Moribund patient not expected to survive > 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Ricordi, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UC-MSCs Group | Control Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UC-MSCs Group | Control Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.58 (15.93) | 58.83 (11.61) | 58.71 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Hemogoblin from Complete Blood Count [Mean (Standard Deviation); unit: g/dL] | 12.93 (2.04) | 12.45 (2.35) | 12.69 (2.17)
Hematocrit from Complete Blood Count [Mean (Standard Deviation); unit: percentage of total blood volume] — Population: Data missing. CBC with differential at baseline was not done in a subset of patients.
  percentage of total blood volume
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 39.71 (6.53) | 40.76 (5.08) | 40.18 (5.79)
White Blood Count (WBC) from Complete Blood Count [Mean (Standard Deviation); unit: 10^3 cells/uL] | 11.87 (5.26) | 14.17 (5.45) | 13.02 (5.37)
Neutrophils from Complete Blood Count [Mean (Standard Deviation); unit: 10^3 cells/uL] — Population: Data missing. CBC with differential at baseline was not done in a subset of patients.
  10^3 cells/uL
    number analyzed (Participants) | 11 | 10 | 21
    (all) | 9.25 (4.8) | 13.37 (5.33) | 11.21 (5.36)
Lymphocytes from Complete Blood Count [Mean (Standard Deviation); unit: 10^3 cells/uL] — Population: Data missing. CBC with differential at baseline was not done in a subset of patients.
  10^3 cells/uL
    number analyzed (Participants) | 11 | 10 | 21
    (all) | 1.15 (0.79) | 0.72 (0.25) | 0.95 (0.62)
Platelet count from Complete Blood Count [Mean (Standard Deviation); unit: 10^3 cells/uL] | 329.83 (99.52) | 342.58 (91.83) | 336.21 (93.88)
Glomerular Filtration Rate from Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 74.5 (31.61) | 61.25 (37.59) | 67.88 (34.63)
Total Protein from Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: g/dL] — Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  g/dL
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 6.39 (0.69) | 6.45 (0.68) | 6.42 (0.67)
Sodium for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mmol/L] | 138.92 (3.15) | 136.58 (5.04) | 137.75 (4.28)
Potassium for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mmol/L] | 4.37 (0.55) | 4.52 (0.67) | 4.44 (0.6)
Creatine for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mg/dL] | 1.18 (0.77) | 1.92 (1.88) | 1.55 (1.46)
Glucose for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mg/dL] | 190.75 (107.14) | 193.67 (85.44) | 192.21 (94.78)
Albumin for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: g/dL] — Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  g/dL
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 3.22 (0.39) | 3.21 (0.51) | 3.22 (0.44)
Alkaline Phosphatase for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: U/L] — Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  U/L
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 90.9 (59.3) | 96.5 (52.69) | 93.7 (54.67)
Alanine Aminotransferase (ALT) or Serum Glutamic-pyruvic Transaminase (SGPT) [Mean (Standard Deviation); unit: U/L] — Alanine Aminotransferase (ALT) or serum glutamic-pyruvic transaminase (SGPT) for comprehensive metabolic panel as assessed from serum blood samples. Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  U/L
    number analyzed (Participants) | 10 | 11 | 21
    (all) | 72.1 (51.19) | 82.45 (75.18) | 77.52 (63.51)
Aspartate Aminotransferase (AST) or Serum Glutamic-Oxaloacetic Transaminase (SGOT) [Mean (Standard Deviation); unit: U/L] — Aspartate Aminotransferase (AST) or Serum Glutamic-Oxaloacetic Transaminase (SGOT) for the comprehensive metabolic panel assessed from serum blood samples. Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  U/L
    number analyzed (Participants) | 10 | 11 | 21
    (all) | 55.8 (31.07) | 118.45 (153.16) | 88.62 (114.86)
Total Bilirubin for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mg/dL] — Population: Data missing. Comprehensive metabolic panel was not completed (only basal metabolic panel) in some patients.
  mg/dL
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 0.62 (0.39) | 0.65 (0.25) | 0.64 (0.32)
Blood Urea Nitrogen (BUN) for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mg/dL] | 29.58 (16.61) | 42.67 (31.27) | 36.13 (25.38)
Calcium for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mg/dL] | 8.53 (0.4) | 8.32 (0.87) | 8.43 (0.67)
Chloride Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mmol/L] | 101 (4.29) | 100.5 (6.33) | 100.75 (5.29)
Carbon Dioxide (CO2) for Comprehensive Metabolic Panel [Mean (Standard Deviation); unit: mmol/L] | 24.42 (3.99) | 21.92 (4.62) | 23.17 (4.41)
Oxygenation Index [Mean (Standard Deviation); unit: Index] — Measure of the fraction of inspired oxygen (FiO2) and its usage within the body during intensive care, measured using fNIRS (Functional Near Infrared Spectroscopy). The calculation for Oxygenation index is ((FIO2 * Mean airway pressure)/partial pressure of oxygen). Population: Data missing. Oxidation Index is only measured and calculated in ventilated patients.
  Index
    number analyzed (Participants) | 4 | 6 | 10
    (all) | 8.09 (2.63) | 14.32 (14.68) | 11.83 (11.5)
Positive End-Expiratory Pressure (PEEP) [Mean (Standard Deviation); unit: cm H2O] — Population: Data missing. PEEP is only measured in patients on ventilator.
  cm H2O
    number analyzed (Participants) | 4 | 7 | 11
    (all) | 13.75 (2.06) | 12.71 (2.14) | 13.09 (2.07)
Plateau Pressure [Mean (Standard Deviation); unit: cm H2O] — Plateau pressure as assessed for patients on a ventilator Population: Data missing. Plateau Pressure is only measured in patients on ventilator.
  cm H2O
    number analyzed (Participants) | 4 | 4 | 8
    (all) | 13.75 (9.74) | 29 (7.39) | 21.38 (11.43)
Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: score on a scale] — Sequential Organ Failure Assessment (SOFA) Scores is used to track a person's risk status during stay in the Intensive Care Unit (ICU). The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each organ system is assigned a point value from a minimum of 0 (normal) to a maximum of 4 (high degree of dysfunction/failure). Totaling a maximum SOFA score of 24 and minimum of 0. Population: Data missing.
  score on a scale
    number analyzed (Participants) | 12 | 11 | 23
    (all) | 5.5 (2.61) | 7.64 (3.35) | 6.52 (3.12)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 97.97 (77.56) | 144.35 (115.69) | 121.16 (99.19)
D-Dimer [Mean (Standard Deviation); unit: mcg/mL FEU] — D-dimer as assessed from serum blood samples. Population: data missing. Collected in a tube that has been recalled by the manufacturer so test was canceled by Quest
  mcg/mL FEU
    number analyzed (Participants) | 12 | 11 | 23
    (all) | 1.76 (2.35) | 4.96 (6.04) | 3.29 (4.69)
Arachidonic Acid/Eicosapentaenoic Acid (AA/EPA) Ratio [Mean (Standard Deviation); unit: ratio of AA to EPA] — ratio of AA to EPA as assessed via serum blood samples.
  ratio of AA to EPA | 45.38 (24.89) | 45.79 (23.93) | 45.58 (23.88)
25-OH vitamin D levels [Mean (Standard Deviation); unit: ng/ml] | 21.76 (8.48) | 23.19 (12.85) | 22.47 (10.68)
Respiratory Rate and Oxygenation Index (ROX) [Mean (Standard Deviation); unit: Index] — The ROX index is the measure of the ratio of pulse oximetry/fraction of inspired oxygen (SpO2/FiO2) to respiratory rate (RR). The ROX index is used as a predictor of the need to intubate in patients receiving HFNC oxygen therapy; performed at 2, 6 and 12 hours. ROX at 2, 6 and 12 hours after HFNC initiation was associated with a lower risk for intubation. For a ROX Index <3.85, risk of HFNC failure is high. If ROX Index 3.85 to <4.88, the scoring could be repeated one or two hours later for further evaluation. Population: data missing. Some patients were on a ventilator. Patients only on HFNC have ROX scores.
  Index
    number analyzed (Participants) | 8 | 5 | 13
    (all) | 7.36 (7.73) | 3.59 (1.13) | 5.91 (6.24)
Viral Load by SARS-CoV-2 RT-PCR [Median (Inter-Quartile Range); unit: copies] — Viral load as assessed in blood plasma for SARS-CoV-2
  copies | 352 [47 to 2184.5] | 3570.50 [175 to 18408.50] | 710 [114 to 10799.50]
Panel Reactive Antibody (PRA) [Count of Participants; unit: Participants] — Panel Reactive Antibody (PRA) for Class I and Class II assessed via serum blood samples
  Participants
    PRA Results Class I: Positive PRA | 11 | 9 | 20
    PRA Results Class I: Negative PRA | 1 | 3 | 4
    PRA Results Class II: Positive PRA | 4 | 6 | 10
    PRA Results Class II: Negative PRA | 8 | 6 | 14
Serology (anti-SARS-CoV-2 IgM and IgG) [Count of Participants; unit: Participants] — Serology (anti-SARS-CoV-2 IgM and IgG) analyzed in blood serum samples. Population: These analyses were implemented in a protocol version that did not apply to two patients of the UC-MSC treatment group and three patients of the control group.
  Participants
    IgM: number analyzed (Participants) | 10 | 9 | 19
    IgM: Positive | 4 | 5 | 9
    IgM: Negative | 6 | 2 | 8
    IgM: Borderline | 0 | 2 | 2
    IgG: number analyzed (Participants) | 10 | 9 | 19
    IgG: Positive | 5 | 8 | 13
    IgG: Negative | 4 | 1 | 5
    IgG: Borderline | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pre-Specified Infusion Associated Adverse Events
Description: Safety as defined by the number of pre-specified infusion associated adverse events as assessed by treating physician. Any of the following occurring within 6 h post each infusion:
  1. An increase in vasopressor dose greater than or equal to the following:
     * Norepinephrine: 10 μg/min
     * Phenylephrine: 100 μg/min
     * Dopamine: 10 μg/kg/min
     * Epinephrine: 10 μg/min
  2. In patients receiving mechanical ventilation: worsening hypoxemia, as assessed by a requirement for an increase of PEEP by 5 cm H2O over baseline, or requirement to increase FiO2 of >20%.
  3. In patients receiving high flow oxygen therapy: worsening hypoxemia, as indicated by requirement of intubation and mechanical ventilation.
  4. New cardiac arrhythmia requiring cardioversion
  5. New ventricular tachycardia, ventricular fibrillation, or asystole
  6. A clinical scenario consistent with transfusion incompatibility or transfusion-related infection
  7. Cardiac arrest or death within 24h post infusion
Time Frame: 6 and 24 hours
Population: In the UC-MSC treatment group, 4 participants were on mechanical ventilation and 8 participants were receiving high flow oxygen therapy. In the control group 7 participants were on mechanical ventilation and 5 participants were receiving high flow oxygen therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Participants
  Number of subjects with an increase in vasopressor dose at 6 h | 1 | 1
  In subjects receiving mechanical ventilation, Number of subjects with worsening of hypoxemia at 6 h: number analyzed (Participants) | 4 | 7
  In subjects receiving mechanical ventilation, Number of subjects with worsening of hypoxemia at 6 h | 1 | 1
  In subjects on high flow oxygen therapy:worsening hypoxemia(req intubat, mechanical ventilat) at 6 h: number analyzed (Participants) | 8 | 5
  In subjects on high flow oxygen therapy:worsening hypoxemia(req intubat, mechanical ventilat) at 6 h | 0 | 0
  Number of subjects with new cardiac arrhythmia requiring cardioversion at 6 h | 0 | 1
  Number of subjects with new ventricular tachycardia, ventricular fibrillation, or asystole at 6 h | 0 | 1
  A clinical scenario consistent with transfusion incompatibility or transfusion-rel infection at 6h | 0 | 0
  Number of subjects with cardiac arrest or death within 24 h post infusion | 0 | 0

2. Primary Outcome: Number of Subjects With Serious Adverse Events by 31 Days After First Infusion
Description: The number of subjects experiencing serious adverse events by 31 days after the first infusion (corresponding to 28 days after the last infusion).
Time Frame: 31 days
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Participants | 2 | 8
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no difference in the number of subjects experiencing serious adverse events in the UC-MSC vs control group"; Test type: Superiority; p = .04, Fisher Exact

3. Primary Outcome: Percentage of Participants Experiencing Serious Adverse Events (SAEs) Through Study Day 90
Description: Safety will be reported as the percentage of participants experiencing serious adverse events through Day 90 as assessed by treating physician.
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
percentage of participants | 41.67 | 66.67

4. Primary Outcome: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Total number of adverse events and serious adverse events as assessed by treating physician
Time Frame: 90 days
Measure: Number; unit: Adverse Events
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Adverse Events
  Number of Adverse Events (not including SAEs) | 40 | 37
  Number of Serious Adverse Events | 6 | 16

5. Primary Outcome: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) by Severity
Description: Total number of adverse events plus serious adverse events categorized by severity.
Time Frame: 90 days
Measure: Number; unit: Adverse Events
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Adverse Events
  Mild | 15 | 13
  Moderate | 22 | 21
  Severe | 9 | 19

6. Primary Outcome: Subjects With Adverse Events and Serious Adverse Events by Severity
Description: Total number of subjects with adverse events and serious adverse events categorized by severity.
Time Frame: 90 days
Population: Subjects who experience one or more AEs or SAEs within each category are counted only once.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Participants
  Mild | 7 | 5
  Moderate | 7 | 8
  Severe | 5 | 7

7. Primary Outcome: Number of Adverse Events and Serious Adverse Events by Relatedness to Treatment
Description: Total number of adverse events and serious adverse events categorized by relatedness to treatment defined by a medical professional.
Time Frame: 90 days
Measure: Number; unit: Adverse Events
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Adverse Events
  Unrelated | 42 | 45
  Unlikely | 3 | 7
  Possible | 1 | 1
  Probably | 0 | 0
  Definite | 0 | 0

8. Primary Outcome: Subjects With Adverse Events by Relatedness to Treatment
Description: Total number of subjects with adverse events categorized by relatedness to treatment by a medical professional
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
Participants
  Unrelated | 8 | 10
  Unlikely | 1 | 4
  Possible | 1 | 1
  Probable | 0 | 0
  Defininte | 0 | 0

9. Secondary Outcome: Survival at 31 Days Post First Infusion
Description: Number of participants that are alive at 31 days post first infusion follow up corresponding to 28 day post second infusion.
Time Frame: 31 Days
Population: One subject in the UC-MSC Group was not included in the data analysis due to failed intubation.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 11 | 12
Participants | 10 | 5

10. Secondary Outcome: Survival at 60 Days Post First Infusion
Description: Number of participants alive at 60 days post first infusion follow up.
Time Frame: 60 days
Population: A subject was censored due to failed intubation in the UC-MSC group.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 11 | 12
Participants | 9 | 5

11. Secondary Outcome: Time to Recovery
Description: Time to discharge or, if the subject was hospitalized, no longer requiring supplemental oxygen and no longer requiring COVID-19-related medical care by 31 days. The numbers represent days at which 25%, 50%, 75% subjects within the treatment group had recovered.
Time Frame: 31 days
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 12
days
  Days by which 75% of subjects were recovered | 23 [13.00 to NA] — insufficient number of people recovered within 31 day limit to estimate the upper confidence | NA [NA to NA] — insufficient number of people recovered within 31 day limit
  Days by which 50% of subjects were recovered | 15 [6 to 23] | NA [10 to NA] — insufficient number of people recovered within 31 day limit
  Days by which 25% of subjects were recovered | 8 [3 to 15] | 12 [9 to NA] — insufficient number of people recovered within 31 day limit to estimate the upper confidence
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no difference in Time to Recovery up to 31 days post infusion between the UC-MSC group and control group". Time to recovery was estimated in each group with Kaplan-Meier survival estimates. Log-rank tests were used to compare hazards between groups; Test type: Superiority; p = 0.0307, Log Rank; Hazard Ratio (HR) = 0.289, 95% CI 2-sided [0.088 to 0.948] — Censoring was limited to dropout from study, and the event of interest was recovery. In the case of death, the patient's time to recovery was censored at the end of study observation; thus the patient remained in the risk set for all KM estimations

12. Secondary Outcome: Ventilator-Free Days Throughout 28 Days Post Second Infusion
Description: Number of days participants were off ventilators during 28 days post second infusion.
Time Frame: 28 days post second infusion
Population: In the UC-MSC treatment group one subject was not included in the analysis due to censoring and another subject was not included due to loss to follow-up. In the control group one subject was not included in the analysis due to discharge against medical advice.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
days | 28 [24 to 28] | 0 [0 to 28]
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; Null Hypothesis: The center of the distributions of ventilator free days are equal in the UC-MSC and control group; Test type: Superiority; p = .0563, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Ventilator-Free Days Throughout 90 Days
Description: Number of days participants were off ventilators within up to 90 days of hospitalization.
Time Frame: 90 days or hospital discharge, whichever is earlier
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
days | 90 [86 to 90] | 0 [0 to 90]
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; Null Hypothesis: The center of the distributions of ventilator free days are equal in the UC-MSC and control group; Test type: Superiority; p = .0563, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Respiratory Rate and Oxygenation Index (ROX Index)
Description: Respiratory Rate-Oxygenation (ROX) index is defined as the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ Fraction of inspired oxygen (FiO2) to respiratory rate. This index can be used in the assessment of disease progression and the risk of intubation in COVID-19 patients with pneumonia.
Time Frame: day 6
Population: ROX index was only measured for patients receiving HFNC and/or not intubated patients. Three patients were ventilated in the UC-MSC group, one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, two patients data was not collected. In the control group one subject was not included in the analysis due to death before day 6, three patients were ventilated, and one patient data was not collected.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 7
Index | 9.57 (5.23) | 7.44 (2.9)

15. Secondary Outcome: Oxygenation Index (OI)
Description: Measure of the fraction of inspired oxygen (FiO2) and its usage within the body during intensive care, measured using fNIRS (Functional Near Infrared Spectroscopy). The calculation for Oxygenation index is ((FIO2 * Mean airway pressure)/partial pressure of oxygen).
Time Frame: day 6
Population: Oxidation Index is only measured and calculated in ventilated patients, therefore 3 patients in the UC-MSC group were included and 3 patients in the control group were included.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 3 | 3
Index | 9.62 (1.43) | 12.74 (5.21)

16. Secondary Outcome: Positive End-Expiratory Pressure (PEEP) and Plateau Pressure (Pplat)
Description: Measuring the respiratory mechanics; positive end-expiratory pressure (PEEP) and plateau pressure (Pplat) in ventilated patients visit 8 (day 6)
Time Frame: day 6
Population: PEEP and Plateau pressure are only measured in ventilated patients, therefore 3 patients in the UC-MSC group were included and 3 patients in the control group were included.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 3 | 3
cm H2O
  PEEP | 9.73 (3.72) | 11.67 (1.53)
  Plateau Pressure: number analyzed (Participants) | 3 | 2
  Plateau Pressure | 28.67 (9.61) | 24 (2.83)

17. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Scores
Description: Sequential Organ Failure Assessment (SOFA) Scores is used to track a person's risk status during stay in the Intensive Care Unit (ICU). The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each organ system is assigned a point value from a minimum of 0 (normal) to a maximum of 4 (high degree of dysfunction/failure). The total score corresponds to the sum of the six different scores of the organ systems. In total, the minimum SOFA score is 0 (normal) and the maximum SOFA score is 24 (highest degree dysfunction/failure).
Time Frame: Day 6
Population: In the UC-MSC treatment group one subject was not included in the analysis due to death and 2 subjects were not included due to discharge on day 6. In the control group one subject was not included in the analysis due to death before day 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 11
score on a scale | 6.56 (2.7) | 6.82 (2.36)

18. Secondary Outcome: Smell Identification Test (SIT) Scores
Description: SIT measures the participant's sense of smell. SIT has a total score ranging from 0 to 40 with the higher the score indicating a more normal sense of smell
Time Frame: 90 days
Population: No participants in the study were able to complete the Smell Evaluation Test due to extenuating circumstances related to the COVID-19 pandemic.
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: White Blood Cell Count (WBC)
Description: As assessed via serum blood samples.
Time Frame: day 6
Population: The UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, and one subject data was not collected. In the control group one subject was not included in the analysis due to death before day 6, two subjects data was not collected.
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
10^3 cells/uL | 13.43 (4.62) | 15.53 (5.6)

20. Secondary Outcome: Platelets Count
Description: As assessed via serum blood samples.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
10^3 cells/uL | 342 (136.33) | 397.89 (135.59)

21. Secondary Outcome: Hemogoblin
Description: Measures the total amount of the oxygen-carrying protein in the blood as assessed via serum blood samples.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
g/dL | 11.93 (2.82) | 11.94 (3.34)

22. Secondary Outcome: Hematocrit
Description: The percentage by volume of red cells in your blood as assessed via serum blood samples.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of red blood cells by volume
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
percentage of red blood cells by volume | 37.98 (8.32) | 36.73 (9.56)

23. Secondary Outcome: Neutrophils
Description: the amount of immune cells (that is one of the first cell types to travel to the site of an infection) as assessed via serum blood samples
Time Frame: day 6
Population: The UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, and two subjects data was not collected. In the control group one subject was not included in the analysis due to death before day 6, two subjects data was not collected.
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 8 | 9
10^3 cells/uL | 9.74 (4.27) | 13.4 (5.95)

24. Secondary Outcome: Lymphocytes
Description: Lymphocyte count as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 8 | 9
10^3 cells/uL | 1.38 (1.07) | 0.8 (0.41)

25. Secondary Outcome: Glomerular Filtration Rate
Description: Glomerular filtration rate (GFR) as assessed via serum blood samples to check how well the kidneys are working. It estimates how much blood passes through the glomeruli each minute.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mL/min/1.73 m^2 | 60.59 (26.99) | 68.67 (35.4)

26. Secondary Outcome: Total Protein
Description: Total protein as assessed via serum blood samples as a part of the comprehensive metabolic panel (CMP). It is a measurement of the sum of albumin and globulins.
Time Frame: Day 6
Population: The UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, and 5 subjects data was not collected. In the control group one subject was not included in the analysis due to death before day 6, and 5 subjects data was not collected.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
g/dL | 5.88 (0.54) | 5.8 (1.06)

27. Secondary Outcome: Sodium
Description: Sodium levels as assessed by serum blood samples.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mmol/L | 141.22 (6.24) | 141 (9.57)

28. Secondary Outcome: Potassium
Description: Potassium levels as assessed via serum blood samples.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mmol/L | 4.25 (0.71) | 4.37 (0.73)

29. Secondary Outcome: Creatinine
Description: Creatinine levels as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mg/dL | 1.21 (0.54) | 1.24 (0.74)

30. Secondary Outcome: Glucose
Description: Glucose levels as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mg/dL | 153.11 (63.99) | 183.89 (82.33)

31. Secondary Outcome: Albumin
Description: Albumin levels as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
g/dL | 2.96 (0.43) | 2.73 (0.45)

32. Secondary Outcome: Alkaline Phosphatase
Description: Alkaline phosphatase levels as assessed via serum blood samples for the Comprehensive Metabolic Panel.
Time Frame: day 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
U/L | 136.2 (68.36) | 202.5 (219.13)

33. Secondary Outcome: Alanine Aminotransferase or Serum Glutamate-pyruvate Transaminase (ALT or SGPT)
Description: The alanine aminotransferase or serum glutamate-pyruvate transaminase (ALT or SGPT) test as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
U/L | 64.4 (38.43) | 65.67 (45.04)

34. Secondary Outcome: Aspartate Aminotransferase or Serum Glutamic Oxaloacetic Transaminase (AST or SGOT)
Description: The aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST or SGOT) test as assessed via serum blood samples
Time Frame: day 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
U/L | 55.8 (23.86) | 47 (32.47)

35. Secondary Outcome: Total Bilirubin
Description: Bilirubin levels as assessed via serum blood samples for the comprehensive metabolic panel.
Time Frame: day 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 6
mg/dL | 0.88 (0.46) | 0.77 (0.29)

36. Secondary Outcome: Blood Urea Nitrogen (BUN)
Description: Blood urea nitrogen (BUN) levels as assessed via serum blood samples for the comprehensive metabolic panel.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mg/dL | 48 (22.28) | 47.67 (26.97)

37. Secondary Outcome: Calcium
Description: Calcium levels as assessed via serum blood samples for the comprehensive metabolic panel.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mg/dL | 8.5 (0.58) | 8.27 (0.67)

38. Secondary Outcome: Chloride
Description: Chloride levels as assessed via serum blood samples for the comprehensive metabolic panel.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mmol/L | 101.56 (7.63) | 102.44 (9.04)

39. Secondary Outcome: Carbon Dioxide (CO2)
Description: Carbon Dioxide (CO2) levels as assessed via serum blood samples for the comprehensive metabolic panel.
Time Frame: day 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 9
mmol/L | 28.44 (3.75) | 26.44 (4.61)

40. Secondary Outcome: C-Reactive Protein Levels
Description: As assessed via serum blood samples.
Time Frame: day 6
Population: In the UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, and data was missing for two subjects. In the control group one subject was not included in the analysis due to death before day 6.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 8 | 11
mg/L | 101.01 (131.05) | 112.55 (104.7)

41. Secondary Outcome: Arachidonic Acid/Eicosapentaenoic Acid (AA/EPA) Ratio
Description: As assessed via serum blood samples on day 6 (visit 8).
Time Frame: day 6
Population: The UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6. In the control group one subject was not included in the analysis due to death before day 6.
Measure: Mean (Standard Deviation); unit: ratio of AA to EPA
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
ratio of AA to EPA | 33.6 (12) | 34.64 (13.24)

42. Secondary Outcome: D-dimer Levels
Description: As assessed via serum blood samples.
Time Frame: day 6
Population: The UC-MSC treatment group one subject was not included in the analysis due to death, one subject was not included due to discharge on day 6, and one subject data was not collected. In the control group one subject was not included in the analysis due to death before day 6 and one subject data was not collected.
Measure: Mean (Standard Deviation); unit: mcg/ml FEU
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 9 | 10
mcg/ml FEU | 6.2 (11.29) | 4.69 (3.38)

43. Secondary Outcome: 25-Hydroxy Vitamin D Levels
Description: As assessed via serum blood samples.
Time Frame: day 6
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
ng/ml | 23.21 (8.91) | 27.58 (16.38)

44. Secondary Outcome: Tumor Necrosis Factor-alpha (TNFα)
Description: Analysis of TNFα in peripheral blood plasma
Time Frame: day 6
Population: In the UC-MSC treatment group one subject was not included in the analysis due to failed intubation. In the control group one subject was not included in the analysis because of death before day 6 blood draw.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 11 | 11
pg/mL | 349 [228 to 407] | 451 [368 to 1730]
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; Test type: Superiority; p = 0.0356, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Tumor Necrosis Factor-beta (TNFβ)
Description: Analysis of TNFβ in peripheral blood plasma
Time Frame: day 6
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 11 | 11
pg/mL | 829 [494 to 1260] | 1540 [852 to 5890]
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; Test type: Superiority; p = 0.0215, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Soluble Tumor Necrosis Factor Receptor 2 (sTNFR2)
Description: Analysis of soluble tumor necrosis factor receptor 2 (sTNFR2) in peripheral blood plasma
Time Frame: day 6
Population: In the UC-MSC treatment group one subject was not included in the analysis due to failed intubation. In the control group one subject was not included in the analysis because of death before day 6 blood draw and data was unavailable for two patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 11 | 9
pg/mL | 26609.09 (3071.96) | 23111.11 (3086.03)
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; Test type: Superiority; p = 0.0210, t-test, 2 sided; Mean Difference (Net) = -3498, 95% CI 2-sided [-6404.7 to -591.2], Standard Deviation 3078.2

47. Secondary Outcome: Viral Load by SARS-CoV-2 RT-PCR
Description: Viral load as assessed in blood plasma for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) via Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).
Time Frame: day 6
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: RNA copies/mL
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
RNA copies/mL | 0 [0 to 0] | 0 [0 to 2193]

48. Secondary Outcome: Number of Participants Reporting Panel Reactive Antibody (PRA) Positivity at Day 3 Post First Infusion
Description: Number of participants reporting panel reactive antibody (PRA) positivity at Day 3 post first infusion for class I and class II as assessed via serum blood samples. These antibodies can develop following a transplant. Recipients can become sensitized to certain molecules (Human Leukocyte Antigen Class I or Class II), which can affect immune responses to and rejection of potential future transplants.
Time Frame: day 3 post first infusion
Population: One subject in the control group died before day 3 post first infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 12 | 11
Participants
  Class I: PRA Positive | 10 | 11
  Class I: PRA Negative | 2 | 0
  Class II: PRA Positive | 4 | 6
  Class II: PRA Negative | 8 | 5
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (class I) status and treatment group at 3 days post first infusion"; Test type: Superiority; p = 0.48, Fisher Exact
Statistical Analysis 2: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (class II) status and treatment group at 3 days post first infusion."; Test type: Superiority; p = 0.41, Fisher Exact

49. Secondary Outcome: Number of Participants Reporting Panel Reactive Antibody (PRA) Positivity at Day 6 Post First Infusion
Description: Number of participants reporting panel reactive antibody (PRA) positivity at Day 6 post first infusion for class I and class II as assessed via serum blood samples. These antibodies can develop following a transplant. Recipients can become sensitized to certain molecules (Human Leukocyte Antigen Class I or Class II), which can affect immune responses to and rejection of potential future transplants.
Time Frame: day 6
Population: In the UC-MSC group one patient was censored and died before day 6 and one patient recovered before day 6 and left the hospital. In the control group on patient died before day 6 post first infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 10 | 11
Participants
  Class I: PRA Positive | 9 | 9
  Class I: PRA Negative | 1 | 2
  Class II: PRA Positive | 5 | 5
  Class II: PRA Negative | 5 | 6
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (class I) status and treatment group at 6 days post first infusion"; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (Class II) status and treatment group at 6 days post first infusion"; Test type: Superiority; p = 1.00, Fisher Exact

50. Secondary Outcome: Number of Participants Reporting Panel Reactive Antibody (PRA) Positivity at Day 14 Post First Infusion
Description: Number of participants reporting panel reactive antibody (PRA) positivity at Day 14 post first infusion for class I and class II as assessed via serum blood samples. These antibodies can develop following a transplant. Recipients can become sensitized to certain molecules (Human Leukocyte Antigen Class I or Class II), which can affect immune responses to and rejection of potential future transplants.
Time Frame: day 14
Population: In the UC-MSC group one patient was censored and died before day 6, 6 patients left the hospital before day 6 post first infusion. In the control group 4 patients died, 3 patients left the hospital and one left hospital against medical advice before day 6 post first infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 5 | 4
Participants
  Class I: PRA Positive | 5 | 3
  Class I: PRA Negative | 0 | 1
  Class II: PRA Positive | 4 | 2
  Class II: PRA Negative | 1 | 2
Statistical Analysis 1: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (class I) status and treatment group at 14 days post first infusion"; Test type: Superiority; p = 0.44, Fisher Exact
Statistical Analysis 2: Comparison: UC-MSCs Group vs Control Group; The null hypothesis is the following: "There is no association between PRA (class II) status and treatment group at 14 days post first infusion"; Test type: Superiority; p = 0.5238, Fisher Exact

51. Secondary Outcome: Number of Participants With Positive, Negative, or Borderline Serology Testing for SARS-CoV-2 IgM/IgG
Description: Number of participants with positive, negative, or borderline SARS-CoV-2 Immunoglobulin M (IgM)/Immunoglobulin G (IgG) serology from serum blood samples.
Time Frame: day 14 post first infusion
Population: These analyses were implemented in a protocol version that did not apply to 2 patients of the UC-MSC treatment group and 3 patients of the control group. In the UC-MSC group one patient was censored and died before day 6, 4 patients left the hospital before day 6 post first infusion and in one patient blood was not drawn. In the control group 3 patients died, 3 patients left the hospital and one left hospital against medical advice before day 6 post first infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | UC-MSCs Group | Control Group
Number analyzed (Participants) | 4 | 2
Participants
  IgM: Positive | 2 | 2
  IgM: Negative | 1 | 0
  IgM: Borderline | 1 | 0
  IgG: Positive | 4 | 2
  IgG: Negative | 0 | 0
  IgG: Borderline | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | UC-MSCs Group | Control Group
All-Cause Mortality (participants affected / at risk) | 3/12 | 7/12
Serious Adverse Events (participants affected / at risk) | 5/12 | 8/12
Other Adverse Events (participants affected / at risk) | 8/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UC-MSCs Group (N=12) | Control Group (N=12)
GI Bleeding 2ry to Clostridium Difficile Infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiact Arrest-Death due to Difficult Intubation (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory Failure 2ry to COVID-Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Death-Acute Hypoxemic Respiratory Failure Secondary to COVID-19 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac Arrest/Pulseless Electrical Activity Cardiac Arrest/Cardiac Arrest Secondary to Acute Respir (Cardiac disorders) | 0 (0) | 3 (3)
Traumatic Tension Pneumotorax post-CPR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
[DEATH] Multisystem Organ Failure (Death)/Multiple Organ Dysfunction Syndrome-Death (General disorders) | 0 (0) | 2 (2)
[DEATH] Cardiac Arrest-Death/Cardiopulmonary Arrest-Death/Asystole -Death (Cardiac disorders) | 1 (1) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Severe Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Septic Shock-Hospital acquired Pseudomona Aeruginosa bacteremia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UC-MSCs Group (N=12) | Control Group (N=12)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Exacerbation of COVID ARDS-Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia after infusion of Investigational Product (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2)
Clostridium Difficile Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mild Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Transaminitis/Transaminitis-Liver Shock (Hepatobiliary disorders) | 0 (0) | 2 (3)
Increased ALT, AST, and Alkaline Phosphatase (Hepatobiliary disorders) | 0 (0) | 1 (1)
Increased Direct Bilirubin (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abnormal Urinalysis (Renal and urinary disorders) | 1 (1) | 0 (0)
Candiduria (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis/Leukocytosis (Increased WBC) (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Severe Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia/Heparin-induced Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bilateral Common Femoral Vein DVT (Vascular disorders) | 0 (0) | 1 (1)
Candida Albicans Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mild Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MRSA Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Paenebacillus Pabuli Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Positive Blood Culture Streptococcus Mitis and Streptococcus Oralis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus haemolyticus bacteremia and Candida orthopsilosi Fungemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcus Hominis Bacteremia/Staphylococcus Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Left Calf Collection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dysconjugated gaze (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute Kidney Injury/Oliguric Acute Kidney Injury/ Anuric Acute Kidney Injury/Acute Kidney Injury (AK (Renal and urinary disorders) | 2 (2) | 5 (5)
Pneumoperitoneum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration Pneumonitis, suspected (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Enterococcus Faecalis, Klebsiella Pneumoniae, Candida Auris/Duobushaemulonis in bronchial aspirate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterococcus Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MRSA Hospital Acquired Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure - Intubation/Hypoxemic respiratory failure requiring intubation and mechanical v (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Subcutaneous Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ventilator Acquired Pneumonia (VAP) with Pseudomona aureginosa (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening of Hypoxemia/Deterioration of Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
The inferences we make from the efficacy results observed in this phase 1/2a trial in 24 subjects, including the outcome of survival, are still subject to limitations of sample size and potential bias because of factors we were not yet aware of.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT04355728/Prot_SAP_000.pdf